CLINICAL TRIAL: NCT04127695
Title: A Randomized, Double-Blind, Placebo Controlled Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of ABBV-0805 in Patients With Parkinson's Disease
Brief Title: A Study to Evaluate the Safety and Tolerability of ABBV-0805 in Patients With Parkinson's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M19-304
Record Dates: First submitted 2019-10-09; First posted 2019-10-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ABBV-0805 Dose 1 or Placebo (Experimental): Participants will receive ABBV-0805 Dose 1 or Placebo.
  Interventions: Drug: ABBV-0805; Drug: Placebo ABBV-0805
- ABBV-0805 Dose 2 or Placebo (Experimental): Participants will receive ABBV-0805 Dose 2 or Placebo.
  Interventions: Drug: ABBV-0805; Drug: Placebo ABBV-0805
- ABBV-0805 Dose 3 or Placebo (Experimental): Participants will receive ABBV-0805 Dose 3 or Placebo.
  Interventions: Drug: ABBV-0805; Drug: Placebo ABBV-0805
- ABBV-0805 Dose 4 or Placebo (Experimental): Participants will receive ABBV-0805 Dose 4 or Placebo. Note: This dosing group may be added after a review of data from dosing groups 1-3.
  Interventions: Drug: ABBV-0805; Drug: Placebo ABBV-0805

INTERVENTIONS:
Drug: ABBV-0805 — ABBV-0805 administered by IV infusion.
Drug: Placebo ABBV-0805 — Placebo ABBV-0805 administered by IV infusion.

SUMMARY:
This study will evaluate the safety and tolerability of ABBV-0805 in adult participants with Parkinson's Disease and results from it will help guide the design of future clinical studies. ABBV-0805 is administered every 28 days by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's Disease (PD) within 5 years and with modified Hoehn and Yahr Stage of less than 3 at Screening.
* Body Mass Index (BMI) is >= 18.0 to <=35.0 kg/m2.
* Participant must follow protocol-specific methods of contraception, if applicable.
* Participant must be in general good health (except for PD) based upon results of medical history, physical examination, vital signs, laboratory testing, neurological examination and 12-lead electrocardiogram (ECG).

Note: If participant is taking standard of care medication for treatment of PD, doses must be stable for at least 30 days prior to starting study drug and participant should not have any clinically relevant motor fluctuations.

Exclusion Criteria:

* Participant with a history of, or screening brain MRI scan indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct > 1 cm3, > 3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space occupying lesion (such as an abscess or brain tumor such as meningioma).
* Received any drug by injection within 30 days or within a period defined by 5 half-lives, whichever is longer, prior to study administration, unless approved by the Investigator in consultation with the AbbVie Therapeutic Area Medical Director.
* Treated with any investigational product within a time frame equal to 5 half-lives, if known, or within 6 weeks (for small molecules) or 6 months (for monoclonal antibodies or other biologics) prior to the first dose of study drug.
* Participant with recent history of drug or alcohol abuse (within 6 months prior to study drug administration) that could impact adherence to the protocol in the opinion of the investigator.
* Participant with evidence of dysplasia or history of malignancy with the exception of excised or treated cervical cancer, some indolent malignancies (such as basal cell carcinoma or squamous cell carcinomas), remission from any malignancy for more than 5 years or participants with slow growth prostatic carcinoma may be eligible to participate with the permission of the AbbVie TA MD.
* Participant with history of seizure disorder or unexplained blackouts or history of a seizure within 6 months.
* Participant with congenital structural or conduction abnormalities, cardiomyopathy, myocardial infarction, cardiac arrhythmias or other cardiac conditions.
* Participant with varicella or herpes zoster virus infection or any severe viral infection within 6 weeks before randomization.
* Received any live vaccine within 4 weeks prior to the first dose of study drug, including but not limited to: measles/mumps/rubella vaccine, varicella zoster virus vaccine, oral polio vaccine, and nasal influenza vaccine.
* Participant with symptoms of an active infection or history of prior infection (viral, fungal, or bacterial) requiring hospitalization or IV antibiotics within 8 weeks before first dose of study drug.
* Participant with history of abnormal laboratory result that, in the opinion of the investigator, are indicative of any significant cardiac, endocrine, hematological, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neurological, and/or other major disease.
* Participant with contraindications to lumbar puncture (such as lumbar scoliosis, coagulopathy, infected skin at needle puncture site). Use of anticoagulants may be allowed in the study but must be temporarily suspended prior to and after lumbar puncture.
* Participant with contraindications to MRI (such as aneurysm clip, metal fragments, internal electrical devices such as a cochlear implant, spinal cord stimulator or pacemaker), are allergic to gadolinium, or have claustrophobia.
* Participant currently enrolled in another interventional clinical study. Participants enrolled in non-interventional studies may be eligible to participate at the discretion of the AbbVie TA MD.
* Participant with clinically significant and/or unstable medical conditions or any other reason that the Investigator determines would interfere with participation in this study or would make the participant an unsuitable candidate to receive ABBV-0805.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Day 1 through Day 260
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Maximum Observed Serum Concentration (Cmax) | Day 1 through Day 29 and Day 85 through Day 113
  Maximum Serum Concentration of ABBV-0805.
Time to Cmax (peak time, Tmax) | Day 1 through Day 29 and Day 85 through Day 113
  Time to Cmax (peak time, Tmax).
Area under the Serum Concentration Time curve (AUC) | Day 1 through Day 29 and Day 85 through Day 113
  Area Under the Serum Concentration Time Curve at first and final dose.
Apparent Terminal Phase Elimination Rate Constant (Beta) | Day 1 through Day 176
  Apparent terminal phase elimination rate constant (Beta) for ABBV-0805.
Ratio of ABBV-0805 concentration in cerebrospinal fluid (CSF) | Day 113
  Concentration of ABBV-0805 in CSF.
Terminal Phase Elimination half-life (t1/2) | Day 1 through Day 176
  Terminal phase elimination half-life (t1/2).
Serum Concentration (Ctrough) | Day 29, Day 57, Day 85, Day 113
  Ctrough concentration of ABBV-0805.
Total clearance (CL) | Day 1 through Day 176
  Clearance of ABBV-0805.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- United States (5):
  - University of Florida - Archer /ID# 212823, Gainesville, Florida
  - Columbia Univ Medical Center /ID# 212826, New York, New York
  - Duke University Medical Center /ID# 214435, Durham, North Carolina
  - Evergreen Neuroscience Institute /ID# 212827, Kirkland, Washington
  - Inland Northwest Research /ID# 212119, Spokane, Washington
- University of Puerto Rico, Medical Sciences Campus /ID# 215751, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: No